CLINICAL TRIAL: NCT00554762
Title: A Phase I, Placebo Controlled, Randomised, Double Blind Two-way Crossover Study to Investigate the Dose Response and Efficacy of Single and Repeat Doses of GW842166 in Healthy Volunteers Using Pharmacodynamic Pain Assessments.
Brief Title: Dose Response and Efficacy of GW842166 in Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Compound terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CBA110877
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Subjects
Keywords: mechanical pain,; heat pain,; dose,; efficacy; dose response,; GW842166,; Single,; pharmacodynamics,; repeat dose,
MeSH Terms: interventions — 2-((2,4-dichlorphenyl)amino)-N-((tetrahydro-2H-pyran-4-yl)methyl)-4-(trifluoromethyl)-5-pyrimidinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW842166X — Administer

SUMMARY:
The purpose of this study is to assess the dose response and efficacy of single and repeat doses of GW842166 in healthy volunteers using pharmacodynamic pain assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 18 to 50 years inclusive
* Body Weight >50 Kg and BMI within the range 18.5 to 32 kg/m2 inclusive.
* Women who are not of child bearing potential

Exclusion Criteria:

* The subject has a positive pre-study urine screen for drugs of abuse or positive alcohol test.
* A positive pre-study (HIV), hepatitis B surface antigen or positive hepatitis C antibody result within 3 months of the start of the study.
* Abuse of alcohol defined as an average weekly intake of greater than 28 units (21 units for women) or an average daily intake of greater than 3 units (2 units for women). 1 unit is equivalent to a half-pint (220 mL) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
• Heat pain threshold at 5 hours post dose | 5 Hours

SECONDARY OUTCOMES:
• Heat pain threshold at 3 hours post dose. • Mechanical pain threshold (using von Frey filaments) at 3 and 5 hours post dose. | 5 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline